CLINICAL TRIAL: NCT01945359
Title: A Pilot Study to Assess Disease State Stability, Efficacy, and Tolerability in a Natalizumab to Dimethyl Fumarate Crossover Design
Brief Title: Pilot Study to Assess Disease Stability in a Natalizumab to Dimethyl Fumarate Crossover Design
Acronym: IIT6
Status: Completed | Type: Observational
Sponsor: Rocky Mountain MS Research Group, LLC (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, John F. Foley, MD, President, Rocky Mountain MS Research Group, Rocky Mountain MS Research Group, LLC
Other Study IDs: 006-001-TEC
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Relapsing Multiple Sclerosis; Dimethyl Fumarate; Natalizumab
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Relapsing Remitting MS (RRMS)

SUMMARY:
This study will observe participants with relapsing remitting multiple sclerosis who are switching therapies from natalizumab to dimethyl fumarate to determine disease stability.

DETAILED DESCRIPTION:
This is an investigator initiated, single site, open-label, single arm observational study examining the initial efficacy and tolerability of dimethyl fumarate in a real world clinical setting for patients with a relapsing form of Multiple Sclerosis (MS) when crossed over from natalizumab therapy.

The decision to cross over from natalizumab to DMF will be made by the patient and the prescribing physician and must precede enrollment in the study.

MS disease status and history will be gathered from the patient's medical records. Patients will be followed for the first 24 weeks of their transition from natalizumab. Assessments will be performed at Baseline and every 4 weeks thereafter for 24 weeks. These assessments may include:

* Expanded Disability Status Scale (EDSS)
* Relapse Assessment
* Patient Reported Outcomes (PRO) including quality of life, fatigue, and cognition outcome measures
* Magnetic Resonance Imaging (MRI)
* Laboratory testing

Study drop outs due to DMF intolerability or other etiologies will be encouraged to complete the trial even if placed on alternative therapies.

ELIGIBILITY:
Inclusion Criteria:

1. JCV Indec of 1.5 of greater and currently receiving natalizumab therapy for at least 24 months
2. Decision to treat with DMF must precede enrollment
3. Ability to understand the purpose and risk of the study and provide authorization for the use of protected health information in accordance with the monitoring agency
4. Men or women >= 18 years at time of informed consent
5. Naive to DMF or fumaric acid esters
6. Confirmed diagnosis of a relapsing form of MS as verified by their treating physician

Exclusion Criteria:

1. Inability ot comply with study requirements as outlined in the informed consent
2. Known active malignancies or any other major co morbidity that, in the opinion of the Investigator, would affect the outcome of the study
3. Pregnancy or breastfeeding
4. Previous treatment with dimethyl fumarate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 participants with relapsing remitting multiple sclerosis crossing over from natalizumab to dimethyl fumarate (DMF) therapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Disease Stability | 8 Months
  Disease stability as measured by stable Expanded Disability Status Scale (EDSS) and no significant changes on magnetic resonance imaging lesions or relapses.

SECONDARY OUTCOMES:
Quantify disease stability | 8 months
  Disease stability will also be assessed by examining annualized relapse rate, proportion of patients experience relapses, Visual Analog Scale (VAS), Modified Fatigue Impact Scale (MFIS), Symbol Digit Modalities Test (SDMT) and pharmacodynamic and pharmacokinetic blood markers.

CONTACTS AND LOCATIONS:
Overall Officials: John F Foley, MD, Principal Investigator — President, Rocky Mountain MS Research Group
Locations (1):
- Rocky Mountain MS Research Group, Salt Lake City, Utah, United States